CLINICAL TRIAL: NCT00610389
Title: Phase II Study With Immunotherapy With Dendritic Cells and Tumor Infiltrating Lymphocytes in Solid Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Ignacio Melero Bermejo, Universidad de Navarra
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD-2007-01
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Last update posted 2010-05-10 (Estimated); Status verified 2010-05

CONDITIONS: Renal Cell Carcinoma; Melanoma; Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Renal Cell; Melanoma; Carcinoma, Hepatocellular | interventions — Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: immunotherapy with dendritic cells

INTERVENTIONS:
Biological: immunotherapy with dendritic cells — We will administer four daily doses (repeated every 24 hours)o dendritic cells in two cycles one month apart. We will administer systemic treatment with PEG-IFN alfa and GM-CSF to potentiate activity.

SUMMARY:
Background: cellular immunotherapy with dendritic cells (DC) loaded with tumor antigens has shown clinical activity, although in a small number of patients. Therefore, is is mandatory to improve the results of this strategy and to closely monitor immunologic response and cell migration in order to improve our understanding of mechanisms of action and to settle future fields of development..

Objectives: Primary: to confirm clinical activity of this strategy, determining tumor response (RECIST criteria). Secondary: to determine: (1) safety; (2) antitumoral immune response and (3) DC migration in the organism

Methodology: phase II trial in patients with advanced renal cell carcinoma and melanoma. We will perform repeated immunizations with DC loaded with the patient´s tumor.

DETAILED DESCRIPTION:
Background: cellular immunotherapy with dendritic cells (DC) loaded with tumor antigens has shown clinical activity, although in a small number of patients. Therefore, is is mandatory to improve the results of this strategy and to closely monitor immunologic response and cell migration in order to improve our understanding of mechanisms of action and to settle future fields of development..

Objectives: Primary: to confirm clinical activity of this strategy, determining tumor response (RECIST criteria). Secondary: to determine: (1) safety; (2) antitumoral immune response (through study of delayed hypersensitivity; ELISPOT; activity of Natural Killer cells; and serum cytokine concentrations); and (3) DC migration in the organism, by labeling with 111-Indium oxinate

Methodology: phase II trial in patients with advanced renal cell carcinoma and melanoma. We will perform repeated immunizations with mature DC loaded with autologous tumor. We will introduce the following novel elements to enhance efficacy (1) Pre-treatment with cyclophosphamide to reduce regulatory / suppressor T cells; (2) maturation/activation of DC induced by TNF-alfa, IFN-alfa and double stranded RNA (GMP-manufactured poly I:C), aimed at replication of the phenomena observed during a viral infection (3) intranodal DC administration in inguinal lymph nodes (4) four daily doses (repeated every 24 hours) in two cycles one month apart (5) scintigraphic follow-up of a tracing dose of 111-In labelled DC and (6) ) systemic treatment with PEG-IFN alfa and GM-CSF to potentiate activity.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of metastatic melanoma, renal cell carcinoma, or hepatocarcinoma (Child´s stage A or B) not amenable of curative treatment. For patients with hepatocarcinoma, treatment after embolization is allowed
* Measurable disease
* ECOG 0, 1 or 2.
* Adequate renal, hepatic and bone marrow function
* Availability of tumor tissue, for maturing dendritic cells

Exclusion Criteria:

* Clinically relevant diseases or infections.
* concurrent participation in other clinical trial or administration or other antitumoral treatment
* Concurrent cancer, with the exceptions allowed by the PI.
* Pregnant or breast feeding women
* immunosuppressant treatment
* known CNS metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2008-02; Primary Completion 2010-04 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Response rate | 2 months

SECONDARY OUTCOMES:
Immunological response | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Melero, MdPhD, Principal Investigator — University of Navarra
Locations (1):
- Oncology Department. Clinica Universitaria de Navarra, Pamplona, Navarre, Spain